CLINICAL TRIAL: NCT00692692
Title: The Use of An Acellular Dermal Matrix Sling in a Two-stage Breast REconstruciton After Mastectomy: A Double-blinded Randomized Trial
Brief Title: Use of Dermal Matrix in Breast Reconstruction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: higher rate of post-operative infection in the Dermal Matrix arm of the study
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 070416
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DermaMatrix (Experimental): experimental group with DermaMatrix acellular dermis over tissue expanders in addition to skin/soft tissue and muscle to allow for more natural appearing breast and prevention of complications
  Interventions: Procedure: DermaMatrix
- Standard of care (Active Comparator): standard of care using skin/soft tissue and muscle coverage of tissue expander for breast reconstruction after mastectomy without acellular dermal matrix
  Interventions: Procedure: standard of care tissue expander breast reconstruction surgery after mastectomy

INTERVENTIONS:
Procedure: DermaMatrix — experimental group with DermaMatrix acellular dermis over tissue expanders in addition to skin/soft tissue and muscle to allow for more natural appearing breast and prevention of complications
  Other Names: tissue expander breast reconstruction after mastectomy
  Arms: DermaMatrix
Procedure: standard of care tissue expander breast reconstruction surgery after mastectomy — standard of care using skin/soft tissue and muscle coverage of tissue expander for breast reconstruction after mastectomy without acellular dermal matrix
  Other Names: standard of care using skin/soft tissue and muscle coverage of tissue expander for breast reconstruction after mastectomy without acellular dermal matrix
  Arms: Standard of care

SUMMARY:
We propose to evaluate the question of whether there is a significant difference between the traditional method of serratus flap tissue expander reconstruction and the acellular matrix method.

DETAILED DESCRIPTION:
We propose a double blinded, randomized study of 60 women comparing outcomes which will include postoperative pain, complication rates and aesthetic outcome as assessed by the patient and a plastic surgeon blinded to the method of reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* All women who are candidates for breast reconstruction using tissue expanders after mastectomy

Exclusion Criteria:

* Other forms of breast reconstruction after mastectomy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wendel, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited from the clinic
Period: Overall Study
Arm/Group | DermaMatrix | Standard of Care
Started | 20 | 16
Completed | 20 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Available data lists demographic data as a single group. Breakdown by arms is not available.
Arm/Group | Both Arms
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction With the Procedure
Time Frame: one year from time of operation
Population: study was terminated and 1 year follow up was not done
Arm/Group | DermaMatrix | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Post Surgical Infection
Description: Number of participants with post surgical infection
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DermaMatrix | Standard of Care
Number analyzed (Participants) | 20 | 16
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | DermaMatrix | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/16
Other Adverse Events (participants affected / at risk) | 6/20 | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DermaMatrix (N=20) | Standard of Care (N=16)
infection (Surgical and medical procedures) | 6 (6) | 2 (2)

LIMITATIONS AND CAVEATS:
Unable to contact PI after he left Vanderbilt. Results were entered with available data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No